CLINICAL TRIAL: NCT00346918
Title: Sirolimus (Rapamune®) for Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD): a Randomized Controlled Study.
Brief Title: Sirolimus (Rapamune®) for Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK-1246
Record Dates: First submitted 2006-06-22; First posted 2006-06-30 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: ADPKD; autosomal dominant polycystic kidney disease; Sirolimus; volumetry
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment of hypertension, cyst infections and flank pain
  Interventions: Other: Standard
- 2 (Active Comparator): Sirolimus plus Standard Treatment
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Standard plus Sirolimus
  Other Names: Rapamune (R)
  Arms: 2
Other: Standard — Standard
  Other Names: Treatment of hypertension, cyst infections and flank pain
  Arms: 1

SUMMARY:
The aim of our study is to investigate whether Rapamune used at a low dose (2 mg/d) retards cyst growth and slows renal functional deterioration in patients with ADPKD.

DETAILED DESCRIPTION:
Currently there is no treatment for ADPKD other than supportive care and blood pressure control. Usually dialytic treatment or renal transplantation becomes necessary when the disease has progressed to end-stage renal failure.We and others could demonstrate that rapamycin, a classical mTOR inhibitor, retards cyst growth and preserves renal function in a rodent model of ADPKD. The aim of our study is to investigate whether Rapamune (2 mg/d) retards cyst growth and slows renal functional deterioration in patients with ADPKD. We anticipate that we can slow disease progression and delay the need for chronic renal replacement therapy by the inhibition of mTOR with Rapamune. This is a 24-month prospective, controlled, open label study with 2 parallel groups in patients with ADPKD. Patients will be randomized at a 1:1 ratio to one of the 2 treatment arms. Primary endpoint is percentage change of renal volume measured by high resolution magnetic resolution imaging.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ADPKD patient between 18 and 40 years of age
* measured GFR higher than 70 ml/min 1.73m2
* documented kidney volume progression
* informed consent

Exclusion Criteria:

* Female of childbearing potential who is planning to become pregnant, who is pregnant and/or lactating, who is unwilling to use effective means of contraception
* increased liver enzymes (2-fold above normal values)
* hypercholesterolemia (fasting cholesterol > 8 mmol/l) or hypertriglyceridaemia (> 5 mmol/l) not controlled by lipid lowering therapy
* granulocytopenia (white blood cell < 3,000/mm3) or thrombocytopenia (platelets < 100,000/mm3),
* infection with hepatitis B or C, HIV
* any past or present malignancy
* mental illness that interfere with the patient ability to comply with the protocol
* drug or alcohol abuse within one year of baseline
* co-medication with strong inhibitor of CYP3A4 and or P-gp like voriconazole, ketoconazole, diltiazem, verapamil, erythromycin
* co-medication with strong CYP3A4 and or P-gp inductor like rifampicin
* known hypersensitivity to macrolides or Rapamune

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2006-06; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
renal volume measured by high resolution magnetic resolution imaging | 1.5 yrs

SECONDARY OUTCOMES:
GFR | 1.5 yrs
Adverse event | 1.5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Andreas L. Serra, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Wahl PR, Serra AL, Le Hir M, Molle KD, Hall MN, Wuthrich RP. Inhibition of mTOR with sirolimus slows disease progression in Han:SPRD rats with autosomal dominant polycystic kidney disease (ADPKD). Nephrol Dial Transplant. 2006 Mar;21(3):598-604. doi: 10.1093/ndt/gfi181. Epub 2005 Oct 12. PMID 16221708
- [Result] Serra AL, Poster D, Kistler AD, Krauer F, Raina S, Young J, Rentsch KM, Spanaus KS, Senn O, Kristanto P, Scheffel H, Weishaupt D, Wuthrich RP. Sirolimus and kidney growth in autosomal dominant polycystic kidney disease. N Engl J Med. 2010 Aug 26;363(9):820-9. doi: 10.1056/NEJMoa0907419. Epub 2010 Jun 26. PMID 20581391
- [Result] Braun M, Young J, Reiner CS, Poster D, Wuthrich RP, Serra AL. Ovarian toxicity from sirolimus. N Engl J Med. 2012 Mar 15;366(11):1062-4. doi: 10.1056/NEJMc1113145. No abstract available. PMID 22417271
- [Result] Braun M, Young J, Reiner CS, Poster D, Krauer F, Kistler AD, Kristanto P, Wang X, Liu Y, Loffing J, Andreisek G, von Eckardstein A, Senn O, Wuthrich RP, Serra AL. Low-dose oral sirolimus and the risk of menstrual-cycle disturbances and ovarian cysts: analysis of the randomized controlled SUISSE ADPKD trial. PLoS One. 2012;7(10):e45868. doi: 10.1371/journal.pone.0045868. Epub 2012 Oct 10. PMID 23071528
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Serra AL, Kistler AD, Poster D, Krauer F, Senn O, Raina S, Pavik I, Rentsch K, Regeniter A, Weishaupt D, Wuthrich RP. Safety and tolerability of sirolimus treatment in patients with autosomal dominant polycystic kidney disease. Nephrol Dial Transplant. 2009 Nov;24(11):3334-42. doi: 10.1093/ndt/gfp280. Epub 2009 Jun 13. PMID 19525519
- [Derived] Serra AL, Kistler AD, Poster D, Struker M, Wuthrich RP, Weishaupt D, Tschirch F. Clinical proof-of-concept trial to assess the therapeutic effect of sirolimus in patients with autosomal dominant polycystic kidney disease: SUISSE ADPKD study. BMC Nephrol. 2007 Sep 15;8:13. doi: 10.1186/1471-2369-8-13. PMID 17868472
- See also: Homepage Study Center — http://www.zystennieren.ch